CLINICAL TRIAL: NCT01587196
Title: CURE Addiction Center of Excellence: Brain Mechanisms of Relapse and Recovery - Prescription Opiates/Medication
Brief Title: CURE Addiction Center of Excellence: Brain Mechanisms of Relapse and Recovery
Acronym: fMRI CURE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 813953
Record Dates: First submitted 2012-04-11; First posted 2012-04-30 (Estimated); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Prescription Opiate/Medication Dependence
Keywords: prescription opiates/medications; vivitrol; brain imaging
MeSH Terms: interventions — vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Naltrexone Intervention (Experimental): Eligible participants receive up to three monthly injections of 380 mg of naltrexone contained in dissolvable polymer microspheres and administered by deep intramuscular injection and slowly released over a period of approximately 4 weeks.
  Interventions: Drug: Vivitrol

INTERVENTIONS:
Drug: Vivitrol — There are monthly injections of depot naltrexone for 3 months.
  Other Names: depot naltrexone (380 mg)

SUMMARY:
The proposed project will use fMRI and specific probes of reward and inhibition as biomarkers predicting drug use during and after treatment in 72 subjects addicted to prescription opioids/medications. Subjects will be scanned before, during, and after 12 weeks of active medication. The brain fMRI measures will be correlated with the primary clinical outcome of drug use (by urine drug screen) during the treatment and follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an informed consent form;
2. Be between the ages of 18 and 60;
3. Have a diagnosis of opioid dependence according to DSM IV-TR criteria (as assessed by the MINI);
4. Be in good general health as determined by complete physical examination and laboratory tests;
5. Have a negative result for urinary opioids and must self report being at least 3 days opioid free. Participants may have a diagnosis of alcohol dependence so long as they do not have severe alcohol dependence that requires medical supervision for alcohol withdrawal.

Exclusion Criteria:

1. Current severe alcohol dependence that requires medical supervision for alcohol withdrawal;
2. Current psychosis, dementia, mental retardation, or history of schizophrenia;
3. Significant clinical abnormalities in hematology, chemistry, or urinalysis;
4. Significant clinical cardiovascular, neurological, hepatic, renal, pulmonary, metabolic, endocrine, or gastrointestinal disorders;
5. Female subjects who are pregnant or lactating, or female subjects of childbearing potential who are not using birth control (oral contraceptives, barrier (diaphragm or condom) plus spermicide, or levonorgestrel implant); (Pregnancy testing will be done on all females of child bearing age); and
6. Current diagnosis of chronic pain disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2012-01; Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Langleben, MD, Principal Investigator — Co-Investigator; Anna R Childress, MD, Principal Investigator — Principal Investigator
Locations (1):
- University of Pennsylvania Addiction Treatment Research Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Wang AL, Shi Z, Elman I, Langleben DD. Reduced cigarette smoking during injectable extended-release naltrexone treatment for opioid use disorder. Am J Drug Alcohol Abuse. 2020 Jul 3;46(4):472-477. doi: 10.1080/00952990.2020.1741001. Epub 2020 May 7. PMID 32379516

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 50 individuals were lost to attrition. 4 individuals withdrew from the study.
Period: Overall Study
Arm/Group | Naltrexone Intervention
Started | 72
Completed | 18
Not Completed | 54
Not completed — Lost to Follow-up | 50
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Naltrexone Intervention
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 72
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 67
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 56
  Race: African American | 11
  Race: American Indian | 0
  Race: Alaskan Native | 0
  Race: Asian/Pacific Islander | 1
  Race: Hispanic (Mexican) | 0
  Race: Hispanic (Puerto Rican) | 3
  Race: Hispanic (Cuban) | 0
  Race: Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Illicit-positive Urines During Treatment and Follow-up
Time Frame: three months
Population: Individuals were tested for presence of opioids: buprenorphine, methadone, opioids, and oxycontin within their urine toxicology
Measure: Count of Participants; unit: Participants
Arm/Group | Naltrexone Intervention
Number analyzed (Participants) | 72
Participants
  Injection One: Buprenorphine | 0
  Injection One: Methadone | 0
  Injection One: Opioids | 1
  Injection One: Oxycontin | 1
  Injection One: Negative Urine Test | 70
  Injection Two: Buprenorphine | 2
  Injection Two: Methadone | 0
  Injection Two: Opioids | 1
  Injection Two: Oxycontin | 2
  Injection Two: Negative Urine Test | 67
  Injection Three: Buprenorphine | 0
  Injection Three: Methadone | 0
  Injection Three: Opioids | 1
  Injection Three: Oxycontin | 0
  Injection Three: Negative Urine Test | 71

ADVERSE EVENTS:
Time Frame: 72 subjects addicted to prescription opioids/medications were scanned before, during, and after 12 weeks of active medication. Participants will receive three injections over three months then be observed for an additional three months
Arm/Group | Naltrexone Intervention
All-Cause Mortality (participants affected / at risk) | 0/72
Serious Adverse Events (participants affected / at risk) | 0/72
Other Adverse Events (participants affected / at risk) | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT01587196/Prot_SAP_000.pdf